CLINICAL TRIAL: NCT02007824
Title: Clinical Trial to Evaluate Efficacy and Safety of Ultrasonic Surgical Device (ULSC-12D)in Chronic Pressure Ulcer
Brief Title: Clinical Trial to Evaluate Ultrasonic Surgical Device in Chronic Pressure Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chan-Yeong Heo, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-2013-020; ULSC-12D (Other: Ultech Ltd.)
Record Dates: First submitted 2013-10-31; First posted 2013-12-11 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Pressure Ulcer; Wound; Necrosis
Keywords: pressure ulcer; chronic wound; tissue necrosis; slough; ultra sound
MeSH Terms: conditions — Pressure Ulcer; Wounds and Injuries; Necrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ULSD-12D (Experimental): ultrasound surgical device made by Ultech.
  Interventions: Device: ULSD-12D
- SONOCA-180 (Active Comparator): ultrasound surgical device made by Soering
  Interventions: Device: SONOCA-180

INTERVENTIONS:
Device: ULSD-12D — wound cleansing and debridement using ULSD-12D
  Arms: ULSD-12D
Device: SONOCA-180 — wound cleansing and debridement using SONOCA-180
  Arms: SONOCA-180

SUMMARY:
Study objective The purpose of this trial is to evaluate the efficacy and safety of the investigational device, ULSD-12D, as Compared to the comparator, SONOCA-180, in chronic wound.

DETAILED DESCRIPTION:
* Study design Multi-center, randomized clinical trial
* Study population Adults with chronic wound
* Investigational device treatment procedure Before Treatment: The subject's eligibility (inclusion/exclusion criteria) will be assessed,and apply the Study Device or Comparator on their wound in a randomized manner. Post-Treatment: All subjects will take pictures of the wound area and measured the number of microorganism and wound size.

ELIGIBILITY:
Inclusion Criteria:

* over 20 years of age
* subject who has untreated wounds
* subject who has wound size over 3cm x 3cm
* subject who has wound over stage 2

Exclusion Criteria:

* cellulitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The number of microorganisms on wound bed | Baseline and 30minuts post debridement
  Investigator measured the number of microorganisms on wound bed at pre and post debridement using nitrocellulose filter.

SECONDARY OUTCOMES:
necrotic tissue region | Baseline and 30minuts post debridement
  Area calculation of necrotic tissue region at pre and post debridement

CONTACTS AND LOCATIONS:
Overall Officials: Chanyeong - Heo, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (3):
- South Korea (3):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Hanyang University Hospital, Seoul, Seongdong-gu